CLINICAL TRIAL: NCT04638010
Title: Increasing Breast, Cervical, and Colorectal Cancer Screening and HPV Vaccination Among Underserved Texans: A Collaboration With the United Way's 2-1-1 Program
Brief Title: Increasing Breast, Cervical, and Colorectal Cancer Screening and HPV Vaccination Among Underserved Texans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Principal Investigator, Maria E Fernandez, Professor and Director, Center for Health Promotion and Prevention Research, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-10-0241
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Cancer Prevention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cancer control navigation (CNN) plus General referral (usual care) (Experimental): Information Specialists at the 2-1-1 call center provide cancer control referrals specific to participant's screening or prevention needs.
  Additionally, Cancer Control Navigators (CNNs) housed at 2-1-1 call centers aid callers. CNNs receive electronic summary profiles of participants assigned to navigation. Navigators call the participant, build a collaborative relationship with them, identify their needs, work with them to identify barriers to services and coordinate solutions, and provide logistic (e.g., making appointments) and emotional support. Navigation services are provided by telephone only.
  Interventions: Behavioral: Cancer control navigation (CNN); Behavioral: General referral (usual care)
- General referral (usual care) (Active Comparator): Information Specialists at the 2-1-1 call center provide cancer control referrals specific to participant's screening or prevention needs.
  Interventions: Behavioral: General referral (usual care)

INTERVENTIONS:
Behavioral: Cancer control navigation (CNN) — Cancer Control Navigators (CNNs) housed at 2-1-1 call centers aid callers. CNNs receive electronic summary profiles of participants assigned to navigation. Navigators call the participant, build a collaborative relationship with them, identify their needs, work with them to identify barriers to services and coordinate solutions, and provide logistic (e.g., making appointments) and emotional support. Navigation services are provided by telephone only.
  Arms: Cancer control navigation (CNN) plus General referral (usual care)
Behavioral: General referral (usual care) — Information Specialists at the 2-1-1 call center provide cancer control referrals specific to participant's screening or prevention needs.

SUMMARY:
This study involves a partnership between UTHealth School of Public Health and the Texas 2-1-1 service, which is a helpline connecting low-income and minority callers with a number of needed services. The purpose of this study is to evaluate the effectiveness of a prevention program in which a phone navigator intervention designed to connect 2-1-1 helpline callers to evidence-based screening and prevention services including mammography, Pap test screening, colorectal cancer screening, and HPV vaccination.

ELIGIBILITY:
Inclusion Criteria:

* callers to 2-1-1
* consents to participate,
* English or Spanish speaking
* not in a crisis (e.g., disaster-related 2-1-1 call or personal crisis)

Exclusion Criteria:

* not English or Spanish speaking
* in crisis (e.g., disaster-related call or personal crisis)
* calling on behalf of another client and not for self

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1554 (Actual)
Dates: Start 2011-02-16 (Actual); Primary Completion 2013-12-06 (Actual); Study Completion 2013-12-06 (Actual)

PRIMARY OUTCOMES:
Number of participants who complete needed cancer screening and prevention services | one month after referral
  Cancer screening and prevention services include mammogram, Pap test, HPV vaccine, and/or colorectal cancer screening.
Number of participants who complete needed cancer screening and prevention services | three months after referral
  Cancer screening and prevention services include mammogram, Pap test, HPV vaccine, and/or colorectal cancer screening.

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Fernandez, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fernandez ME, Savas LS, Atkinson JS, Ricks KB, Ibekwe LN, Jackson I, Castle PE, Jobe D, Vernon SW. Evaluation of a 2-1-1 Telephone Navigation Program to Increase Cancer Control Behaviors: Results From a Randomized Controlled Trial. Am J Health Promot. 2022 Sep;36(7):1083-1093. doi: 10.1177/08901171211041276. Epub 2022 May 5. PMID 35514063